CLINICAL TRIAL: NCT05119244
Title: Environment and Lung Cancer
Acronym: PPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021-A02062-39
Record Dates: First submitted 2021-11-02; First posted 2021-11-15 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Cannabis Use
Keywords: Cannabis, Lung Cancer
MeSH Terms: conditions — Marijuana Abuse; Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- cannabis smokers (Experimental)
  Interventions: Other: blood and hair sampling
- Tobacco smokers (Experimental)
  Interventions: Other: blood and hair sampling
- Non-smoking patients (Experimental)
  Interventions: Other: blood and hair sampling

INTERVENTIONS:
Other: blood and hair sampling — 3.5 ml blood sample Hair sample

SUMMARY:
Cannabis is the most consumed drug in the world and the French are the main consumers in Europe. The most recognized effects of cannabis on human health are of a neuro-psychic nature. The medical literature on the effects of cannabis on the lung in general, and on lung carcinogenesis in particular, is most often reassuring (Tashkin, Chest 2018; Zhang, Int J Cancer 2015; Ghasemiesfe JAMA Netw. Open. 2019), despite the fact that the concentration of carcinogens in cannabis smoke is higher than that contained in tobacco smoke (Moir, Chem. Res. Toxicol. 2008), and that cannabis smoking has been implicated in the occurrence of ENT cancers. Rather, research focuses on the therapeutic effects of cannabis, especially analgesics, and even on its possible anti-tumor virtues (Abrams, Jama Oncol. 2020). These reassuring data should, however, be viewed with a great deal of caution. On the one hand, the illegal nature of cannabis in most countries and its frequent association with tobacco consumption make studies on the subject difficult and often biased. On the other hand, the daily practice of oncologists, who observe numerous cases of advanced and rapidly progressive lung cancer occurring in young patients who are heavy users of cannabis, raises suspicion of an unrecognized role of cannabis in lung carcinogenesis.

In a preliminary multicenter study on French patients under 50 years of age operated for primary lung cancer (Betser, ERJ 2021), we demonstrated that cannabis consumption was extremely frequent, concerning 43% of patients, but mentioned in patients' medical records only in 4 out of 10 cases, while the smoking status was always noted.

In addition, by comparing people who smoke cannabis (always here associated with tobacco) to patients who only smoke tobacco or to non-smokers, we identified a different profile of lung cancers, with more poorly differentiated tumors, presenting at a more advanced stage (more T3-T4 versus T1-T2) requiring more complex surgery, and mostly located in the upper lobes of the lung.

Similar research work is currently underway at Gustave Roussy (Dr Pradere-Dr Planchard, Villejuif, France) on patients with metastatic lung cancer, with a focus on overall survival and molecular profile.

ELIGIBILITY:
Inclusion Criteria:

* Any patient from 18 y.o to 59 y.o treated in one of the three above-mentioned hospitals for primary lung cancer, whatever its stage, and agreeing to participate in this research.

Exclusion Criteria:

* Patient denied participation.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
percentage of patients who are active or not active cannabis smokers (at least 10 joints per for at least one year). | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson
  - Institut Gustave Roussy, Villejuif